CLINICAL TRIAL: NCT01401712
Title: Thoracic Epidural Analgesia Compared to Thoracic Paravertebral Pump Infusion for Pain Management in Patients With Three or More Rib Fractures
Brief Title: Optimal Method of Pain Management in Patients With Multiple Rib Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: I-Flow (Industry)
Responsible Party: Principal Investigator, George Velmahos, Division Chief, Trauma, Emergency Surgery, Surgical Critical Care, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011P001678
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: 3 or More Rib Fractures
Keywords: ON-Q; epidural; analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paravertebral catheter (ON-Q® Pain Relief System) (Experimental)
  Interventions: Procedure: ON-Q® Pain Relief System
- Thoracic epidural catheter (Active Comparator)
  Interventions: Procedure: Thoracic epidural catheter

INTERVENTIONS:
Procedure: ON-Q® Pain Relief System — Identify insertion site lateral to paraspinous muscles and posteromedial to the rib fractures. Then, incise skin and soft tissue down to the level of the rib. Advance tunneler perpendicular to chest wall until it contacts the rib, then, advance superiorly at 45° angle in the extrathoracic space. Remove tunneler and advance catheter in space created. Attach catheter to pump filled with 0.2% ropivacaine at infusion rate of 2-12ml/hr.
  Arms: Paravertebral catheter (ON-Q® Pain Relief System)
Procedure: Thoracic epidural catheter — Introduce needle into the interspinous space of the vertebral column and advance into the epidural space. Advance the epidural catheter about 3-5 cm into the epidural space and remove the needle.
  Arms: Thoracic epidural catheter

SUMMARY:
Rib fractures are a common injury of trauma patients and can cause significant pain which, if inadequately treated, can lead to impaired breathing, lung collapse, and respiratory failure. Hence, it is crucial to manage pain associated with rib fractures. Currently, epidurals are used to treat the pain, but placement can be risky as rib fractures are often associated with other injuries and complications.

An alternative pain management option is the ON-Q® Pain Relief System. It is an FDA-approved device that automatically and continuously delivers medication to the region of the thoracic intercostal nerves. One study by Truitt et al (2010)demonstrated that the ON-Q® system effectively reduced pain and increased lung volumes after one hour, in patients with three or more rib fractures. However, that study sample was small and did not have a comparison group. In this study, we will compare two groups: 1) ON-Q system and 2) epidural analgesia. We hypothesize that trauma patients with three or more rib fractures, who receive pain management through the ON-Q® Pain Relief System achieve discharge criteria earlier and thus have a shorter hospital length of stay (LOS) when compared with epidural analgesia.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years;
2. Three or more rib fractures;
3. Pain

   1. Severe pain (i.e. causing deleterious affect on respiratory mechanics, respiratory rate, or oxygen saturations), OR
   2. Mild to moderate pain (i.e. minimally affecting respiratory mechanics, respiratory rate, or oxygen saturations) that does not respond to oral or intravenous analgesics within 4 hours;
4. Patient has capacity to provide informed consent, as determined by:

   1. Clinical assessment by study staff MD who will explain the study to potential subjects and then ask them to summarize the purpose, procedures, risks and alternatives back to the MD;
   2. GCS 15;
   3. Clinical assessment by independent MD who will explain the study to potential subjects and then ask them to summarize the purpose, procedures, risks and alternatives back to the MD.

Exclusion criteria:

1. Lack capacity to provide informed consent;
2. Intubation at time of enrollment;
3. Contraindications to procedure (e.g. known allergy to local anesthetics).
4. Presence of infection at site of catheter placement;
5. Current use of anticoagulant medication;
6. Known allergy to silver;
7. Inability to obtain informed consent;
8. Body weight > 300 lbs;
9. Pregnancy;
10. Significant co-morbid medical illness that might alter the metabolism of the anesthetic agents and result in unexpected toxicity (hepatic, renal or cardiopulmonary disease).

All women of child-bearing age will receive a urine pregnancy test prior to the start of the interventional portion of the study. A positive test result excludes the patient from inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay/time to achieve discharge criteria | Patient will be followed for the duration of hospital stay, 1 week
  The study will compare the time to achieve discharge criteria between the two groups. Readiness for discharge is defined by the following criteria:
  1. Visual Analog Score (VAS) for pain below 4 (of a maximum 10);
  2. Ability to perform incentive spirometry with sustained maximal inspiration for three seconds;
  3. Hemodynamic stability (heart rate <100 beats/min, respiratory rate <20 breaths/min, and systolic blood pressure >90mmHg at 3 consecutive time points that are 10 minutes apart) and oxygen saturation greater than 95% on room air;
  4. Absence of neurological deficits; and
  5. Monitored for at least 1 hour after ON Q® catheter placement to ensure no immediate complications from placement or local anesthestic toxicity.

SECONDARY OUTCOMES:
Pain score reduction | Patient will be followed for duration of hospital stay and through daily phone calls upon discharge
  Decrease in pain as measured by the Visual Analog Scale (VAS) pre-placement and 60 min post-placement of intervention. Pain score will be followed for the duration of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: George C Velmahos, Md, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Truitt MS, Mooty RC, Amos J, Lorenzo M, Mangram A, Dunn E. Out with the old, in with the new: a novel approach to treating pain associated with rib fractures. World J Surg. 2010 Oct;34(10):2359-62. doi: 10.1007/s00268-010-0651-9. PMID 20567973